CLINICAL TRIAL: NCT06292832
Title: Ultrasound-guided Erector Spinae Plane Block Versus Transversus Abdominis Plane Block for Pain Control After Cesarean Section in Obese and Morbidly Obese Women
Brief Title: Erector Spinae Plane Versus Transversus Abdominis Plane Block for Pain Control
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Warda Demerdash Khalifa Ali, Principal investigator, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MSR/AZAST/AIP029/22/222/8/2023
Record Dates: First submitted 2024-02-20; First posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-02

CONDITIONS: Cesarean Section Complications

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Obese Spinae Plane Block (Active Comparator): Spinae Plane Block for pain control
  Interventions: Procedure: Ultrasound-guided pain block; Device: Ultrasound Machine
- Obese Transversus Abdominis Plane Block (Active Comparator): Transversus Abdominis Plane Block for pain control.
  Interventions: Procedure: Ultrasound-guided pain block; Device: Ultrasound Machine
- Morbidly Obese Spinae Plane Block (Active Comparator): Spinae Plane Block for pain control
  Interventions: Procedure: Ultrasound-guided pain block; Device: Ultrasound Machine
- Morbidly Obese Transversus Abdominis Plane Block (Active Comparator): Transversus Abdominis Plane Block for pain control.
  Interventions: Procedure: Ultrasound-guided pain block; Device: Ultrasound Machine

INTERVENTIONS:
Procedure: Ultrasound-guided pain block — Ultrasound-guided pain block after cesarean section
Device: Ultrasound Machine — Ultrasound machine used to guide the nerve block.

SUMMARY:
The present stratified randomized study aimed to compare the analgesic efficacy and safety profile of ESPB and TAPB used for postoperative pain management in obese and morbidly obese women undergoing CS.

DETAILED DESCRIPTION:
The present stratified randomized study aimed to compare the analgesic efficacy and safety profile of ESPB and TAPB used for postoperative pain management in obese and morbidly obese women undergoing CS. The present study will include ASA I-II women scheduled for elective CS under intrathecal anesthesia. Patients will be excluded if they had local infection, bleeding disorder or known allergy to any of the study medications. This study defines obesity as body mass index (BMI) ≥ 30 kg/m2 while morbid obesity is defined as BMI ≥ 40 kg/m2 assessed in the last pre-pregnancy visit (Sagi-Dain et al., 2021). The study will include normal weight women (n=86), obese women (n=86) and morbidly obese women (n=86).

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II women scheduled for elective CS under intrathecal anesthesia.

Exclusion Criteria:

* had local infection, bleeding disorder or known allergy to any of the study medications

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2024-03-10 (Estimated); Primary Completion 2024-09-10 (Estimated); Study Completion 2024-09-10 (Estimated)

PRIMARY OUTCOMES:
postoperative time to rescue analgesia requirement | 24 hours
  Time

CONTACTS AND LOCATIONS:
Overall Officials: Warda Ali, Principal Investigator — Al-Azhar University, Assiut, Egypt
Locations (1):
- Al-Azhar University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No